CLINICAL TRIAL: NCT04491201
Title: National Survey of the Impact of COVID-19 Pandemics on Chinese Physicians of Obstetrics and Gynecology
Brief Title: National Survey of the Impact of COVID-19 Pandemics
Acronym: CMDA-SURVEY2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CMDA-SURVEY2
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: COVID-19 Pandemics; Obstetrics and Gynecology; Workload; Questionnaire; National Survey; China
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Customized questionnaire — A customized questionnaire will be delivered by the social software WeChat to the specific hospital which has been randomly sampled, and all physicians of Obstetrics and Gynecology in this hospital will fill the questionnaire anonymously.

SUMMARY:
COVID-19 pandemics have changed extensively the lives around the world. Although most physicians of obstetrics and gynecology have no critical role in the frontline against COVID-19 pandemics, their work, research and education activities still underwent great changes. The primary aim of this study is to analyze change of workload during the COVID-19 pandemics in physicians of obstetrics and gynecology in China. A customized questionnaire will be delivered by the social software WeChat to the specific hospital which has been randomly sampled, and all physicians of Obstetrics and Gynecology in this hospital will fill the questionnaire anonymously.

A random sampling will be performed in all 32 provinces, municipality or autonomous regions in the mainland of China. It is assumed that acceptable 95% confidence interval is P±4%, and the sample size under the condition of simple random sampling is 600 persons. If the homogeneity is set as 0.15 or 0.2, and each population (unit) has 10 or 15 persons accepting survey, we will achieve a design effect of 2.35 to 3.80. If we choose the design effect of 3, the sample size of every level needs is 1800. Considering 10% population refusing to be surveyed, in all mainland of China, three levels of hospitals will include at least 6000 physicians who accept survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old
* Belonging to and registered at specific hospital
* Active employment in obstetrics, reproduction, or gynecology
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all the inclusion criteria
* Not completing the whole questionnaire

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All physicians of obstetrics and gynecology from the hospitals randomly sampled
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-27 (Estimated); Study Completion 2020-09-27 (Estimated)

PRIMARY OUTCOMES:
The changes of workload of physicians during COVID-19 pandemics compared with 2019 year | Six months
  Reduction or augment in percentage of workload including outpatient clinics, surgeries, counseling and deliveries

SECONDARY OUTCOMES:
The changes of education activities during COVID-19 pandemics compared with 2019 year | Six months
  Reduction or augment in percentage of education activities including lectures, ward rounds and exams.
The changes of research activities during COVID-19 pandemics compared with 2019 year | Six months
  Reduction or augment in percentage of research activities including research protocol advancement, paper composition/submission/publication, and fund application

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li L, Cao Y, Fan J, Li T, Lang J, Zhang H, Lv J, Zhu L; Chinese Medical Doctor Association. Impact of COVID-19 Pandemic on the Clinical Activities in Obstetrics and Gynecology: A National Survey in China. Front Med (Lausanne). 2021 Jul 30;8:633477. doi: 10.3389/fmed.2021.633477. eCollection 2021. PMID 34395457